CLINICAL TRIAL: NCT00392912
Title: A Pilot Study of the Effect of Testosterone on Cerebral Glucose Metabolism in Hypogonadal Males With Alzheimer's Disease
Brief Title: Effect of Testosterone Therapy in Men With Alzheimer's Disease and Low Testosterone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michael E. DeBakey VA Medical Center (U.S. Federal Agency)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Robert Tan, MD
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GR-294
Record Dates: First submitted 2006-10-24; First posted 2006-10-26 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Alzheimer's Disease; Hypogonadism
Keywords: testosterone; hypogonadal; cerebral glucose metabolism; PET scan; Alzheimer's disease
MeSH Terms: conditions — Alzheimer Disease; Hypogonadism | interventions — Testosterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AndroGel (Solvay Pharmaceuticals) — Testosterone Replacement Therapy: AndroGel 1% 5g packets (Solvay Pharmaceuticals). Initial dosage: 5g daily (1 packet). Patients who do not achieve eugonadal levels of 400-600 mg/dL within 2 weeks will be raised to 10g daily.
  Other Names: AndroGel 1% 5g packets (Solvay Pharmaceuticals)

SUMMARY:
Treatment with testosterone can improve performance on tests of spatial ability in men with low testosterone levels and Alzheimer's disease. Improved performance on these tests may mean an improved ability to get around in one's environment without getting lost or injured. This could have a positive impact on both patients and those who care for them. We will investigate what areas of the brain are involved in these improvements in spatial ability. This will be done using a PET scan, which creates a 3-dimensional image of the brain that can allow us to see how the brain functions.

DETAILED DESCRIPTION:
Volunteers will be treated with a prescription testosterone gel applied to the shoulder or other body area each day. This treatment will continue for 6 months. Subjects will undergo a PET scan at the beginning of the study and after approximately 2 months of treatment. Subjects will undergo some cognitive testing throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Alzheimer's disease diagnosis, based on Diagnostic and Statistical Manual of Mental Disorders (5th ed.; DSM-V)
* Total testosterone < 300 ng/dL and/or calculated free testosterone < 50 pg/ml
* Sufficient English to perform cognitive testing
* Stable on concomitant medications for 1 month prior to starting study

Exclusion Criteria:

* history of prostate cancer
* history of breast cancer
* gonadal endocrine disorders
* current major psychiatric illness (excluding depression)
* significant uncontrolled systemic illness
* recent myocardial infarction (within 6 months)
* renal or hepatic disease, sleep apnea
* history of alcoholism or substance abuse within the past year
* history of head injury with loss of consciousness greater than 1 hour
* testosterone or other androgen treatment within past 3 months
* history of taking other drugs that might interfere with the results of the study (ie, spironolactone, cimetidine, antiandrogens, estrogens, p450 enzyme inducers, barbiturates)
* symptomatic BPH: prostatic symptoms, prostatic masses or induration on rectal examination
* prostate specific antigen (PSA) >4.0 mg/mL
* hemoglobin > 17 mg/dL
* generalized skin disease that could affect the absorption of testosterone gel (ie, psoriasis).
* potentially agitated or uncooperative for procedures

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2007-04; Primary Completion 2009-11 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Calculated difference image of pre-treatment and on-treatment PET scans.

SECONDARY OUTCOMES:
Change in cognitive function at 8-week intervals over a 6-month period.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tan, MD, Principal Investigator — Michael E. DeBakey VA Medical Center, Houston, TX
Locations (1):
- Michael E. DeBakey VA Medical Center, Houston, Texas, United States